CLINICAL TRIAL: NCT06132113
Title: DAREON™-7: A Phase I, Open-label, Dose Escalation and Expansion Trial to Investigate Safety and Tolerability of BI 764532 Intravenous Infusions in Combination With Standard of Care (Platinum and Etoposide) in First-line Treatment of Patients With Neuroendocrine Carcinomas (NEC)
Brief Title: DAREON™-7: A Study to Test How Well Different Doses of BI 764532 in Addition to Chemotherapy Are Tolerated by People With Advanced Neuroendocrine Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1438-0007; U1111-1292-1400 (Registry Identifier: WHO Registry); 2023-505870-13-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Neuroendocrine Neoplasms
MeSH Terms: interventions — Carboplatin; Etoposide; Cisplatin

STUDY DESIGN:
Intervention Model Description: Part A1: Dose escalation, Part A2: Reduced monitoring, Part B: Dose expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A1: BI 764532 low dose + carboplatin + etoposide (Experimental)
  Interventions: Drug: BI 764532; Drug: Carboplatin; Drug: Etoposide
- Part A1: BI 764532 medium dose + carboplatin + etoposide (Experimental)
  Interventions: Drug: BI 764532; Drug: Carboplatin; Drug: Etoposide
- Part A1: BI 764532 high dose + carboplatin + etoposide (Experimental)
  Interventions: Drug: BI 764532; Drug: Carboplatin; Drug: Etoposide
- Part B: BI 764532 + carboplatin + etoposide (Experimental)
  Interventions: Drug: BI 764532; Drug: Carboplatin; Drug: Etoposide
- Part B: BI 764532 + cisplatin + etoposide (Experimental)
  Interventions: Drug: BI 764532; Drug: Etoposide; Drug: Cisplatin
- Part A2: BI 764532 + carboplatin + etoposide (Experimental)
  Interventions: Drug: BI 764532; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: BI 764532 — BI 764532
  Other Names: Obrixtamig
Drug: Carboplatin — Standard of care
  Arms: Part A1: BI 764532 high dose + carboplatin + etoposide; Part A1: BI 764532 low dose + carboplatin + etoposide; Part A1: BI 764532 medium dose + carboplatin + etoposide; Part A2: BI 764532 + carboplatin + etoposide; Part B: BI 764532 + carboplatin + etoposide
Drug: Etoposide — Standard of care
Drug: Cisplatin — Standard of care
  Arms: Part B: BI 764532 + cisplatin + etoposide

SUMMARY:
This study is open to adults aged 18 and older or above legal age who have a specific type of advanced neuroendocrine cancer (NEC). Their tumours must be positive for a marker called DLL3.

The purpose of this study is to test a medicine called BI 764532 in addition to chemotherapy. The study has Part A1, Part A2, and Part B. Part A1 of this study aims to find out the highest dose of BI 764532 that people can tolerate in addition to chemotherapy. Part A2 of this study is to find out how well people tolerate a low dose of BI 764532 combined with the chemotherapy. The purpose of Part B is to find out how well people can tolerate BI 764532 in combination with different chemotherapies. Researchers also want to find out whether BI 764532 in combination with chemotherapy helps people with NEC.

Participants get different doses of BI 764532 as an infusion into a vein. In addition, they get platinum-based chemotherapy as infusions into a vein. Participants can continue treatment up to 3 years if they benefit from treatment and can tolerate it.

Participants visit their doctors regularly. During these visits, the doctors collect information about participants' health and take note of any unwanted effects. Doctors also regularly check the size of the tumour.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants ≥18 years old and at least at the legal age of consent in countries where it is greater than 18 years at the time of signature of the informed consent form (ICF)
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to any trial-specific procedures, sampling, or analyses
* Patients diagnosed with locally advanced or metastatic NEC of following subtypes:

  * extrapulmonary neuroendocrine carcinomas (epNEC)
  * pulmonary large cell NEC (LCNEC)
  * neuroendocrine carcinomas (NEC) of unknown primary site
* Patients with tumours with mixed histologies for any above type are eligible only if neuroendocrine carcinoma/small tumour cells component is predominant and represent at least 50% of the overall tumour tissue
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Minimum life expectancy of 12 weeks
* At least one measurable lesion as defined per RECIST 1.1 within approximately 35 days prior to the first dose of BI 764532
* Patients with a history of asymptomatic Central nervous system (CNS) metastases are eligible, provided they meet all of the following criteria:

  * No radiotherapy (including whole brain radiation therapy, stereotactic radiotherapy or radiosurgery) within 7 days
  * Are neurologically stable without the need for steroids or anti-convulsants for at least 7 days before first dose of BI 764532 as per local site assessment Further inclusion criteria apply.

Exclusion Criteria:

* Previous treatment in this trial
* Current enrolment in another investigational device or drug trial, or <30 days since ending another investigational device or drug trial(s)
* Patients with diagnosis of Merkel cell carcinoma or medullary thyroid carcinoma or Grade 3 neuroendocrine tumour
* Presence of leptomeningeal carcinomatosis
* Previous treatment with DLL3-targeting T cell engagers and cell therapies
* Patients who have been treated with extensive field radiotherapy including whole brain irradiation within 2 weeks prior to first administration of BI 764532
* Major surgery (major according to the investigator's assessment) within 28 days prior to first administration of BI 764532 or planned during treatment period, e.g. hip replacement Any documented active or suspected malignancy or history of malignancy within 5 years prior to Screening (other than the target indication or well differentiated neuroendocrine tumour (NET) stages of the target indication in case of transformed tumors), except for appropriately treated basal cell carcinoma of the skin or in situ carcinoma of uterine cervix Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2027-02-09 (Estimated); Study Completion 2027-04-25 (Estimated)

PRIMARY OUTCOMES:
Part A1: Occurrence of dose-limiting toxicities (DLTs) in the maximum tolerated dose (MTD) evaluation period | Up to 21 days.
Part A2: Reduced monitoring: the occurrence of DLTs during the on-treatment period | Up to 36 months.
Part B: Occurrence of dose-limiting toxicities (DLTs) during the on-treatment period | Up to 36 months.

SECONDARY OUTCOMES:
Part A1: Occurrence of dose-limiting toxicities (DLTs) during the on-treatment period | Up to 36 months.
Part A1: Occurrence of adverse events (AEs) during the on-treatment period | Up to 36 months.
Part A2: Occurrence of adverse events (AEs) during the on-treatment period | Up to 36 months.
Part A2: Objective response (OR) | Up to 36 months.
  Objective response (OR), defined as a best overall response of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST 1.1 (based on investigator's assessment) from the date of treatment start until the earliest date of disease progression, death, or last evaluable tumour assessment before start of subsequent anti-cancer therapy, loss to follow-up, or withdrawal of consent.
Part B: Objective response (OR) | Up to 36 months.
  Objective response (OR), defined as a best overall response of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST 1.1 (based on investigator's assessment) from the date of treatment start until the earliest date of disease progression, death, or last evaluable tumour assessment before start of subsequent anti-cancer therapy, loss to follow-up, or withdrawal of consent.
Part B: Duration of response (DoR) | Up to 36 months.
  Duration of response (DoR), defined as the time from first documented confirmed objective response (OR) until the earliest date of disease progression or death among patients with confirmed objective response.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (5):
  - University of Miami, Miami, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - John Theurer Cancer Center, Hackensack, New Jersey
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- France (2):
  - HOP Louis Pradel, Bron
  - INS Paoli-Calmettes, Marseille
- Germany (2):
  - Klinikum der Universität München AÖR, München
  - Universitätsklinikum Tübingen, Tübingen
- Japan (4):
  - Aichi Cancer Center Hospital, Aichi, Nagoya
  - National Cancer Center Hospital East, Chiba, Kashiwa
  - Osaka International Cancer Institute, Osaka, Osaka
  - National Cancer Center Hospital, Tokyo, Chuo-ku
- Universitair Medisch Centrum Groningen, Groningen, Netherlands
- Spain (3):
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
- Sweden (2):
  - Sahlgrenska Universitetsjukhuset, Gothenburg
  - Akademiska hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com